CLINICAL TRIAL: NCT01311466
Title: Open Non-randomized Study to Assess the Benefit of Liver Transplantation in Patients With Liver Metastasis After Ocular Malignant Melanoma (Uveal Melanoma)
Brief Title: Liver Transplantation and Uveal Malignant Melanoma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oslo University Hospital (Other)
Responsible Party: Principal Investigator, Svein Dueland, MD PhD, Oslo University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: S-06408
Record Dates: First submitted 2011-03-07; First posted 2011-03-09 (Estimated); Last update posted 2017-10-23 (Actual); Status verified 2017-10

CONDITIONS: Uveal Malignant Melanoma
Keywords: Liver transplantation; Overall survival
MeSH Terms: interventions — Liver Transplantation

ARMS (1):
- Liver transplantation (Experimental): The liver transplantation will be performed as described by the standard protocol, Liver Transplantation Protocol (Version 2006) at the Oslo University Hospital
  Interventions: Procedure: Liver transplantation

INTERVENTIONS:
Procedure: Liver transplantation

SUMMARY:
Patients with uveal malignant melanoma with liver metastases have median survival of less than 12 months. There is no established treatment showing increased overall survival. The study will determine if liver transplantation will result in long term survival in patients with liver metastases from uveal malignant melanoma.

ELIGIBILITY:
Inclusion Criteria:

* Uveal malignant melanoma
* Liver metastases
* ECOG 0-1

Exclusion Criteria:

* Extra hepatic disease
* Previous other malignancy
* Previous organ transplantation

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2011-01; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Over all survival | 1 year
  Patient survival after livertransplantation

CONTACTS AND LOCATIONS:
Overall Officials: Svein Dueland, MD, PhD, Principal Investigator — Oslo University Hospital, Radium hospitalet
Locations (1):
- Oslo University Hospital, Oslo, Norway